CLINICAL TRIAL: NCT06548490
Title: GLP-1R Agonist Treatment for Opioid Use Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: New York University (Other); University of Maryland (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Patricia Sue Grigson, Chairperson (Academic Administrator) Neural and Behavioral Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00024676; UH3DA050325 (NIH)
Record Dates: First submitted 2024-08-07; First posted 2024-08-12 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Opioid Use Disorder; Opioid Abuse and Addiction; Narcotic-Related Disorders; Substance-Related Disorders; Chemically-Induced Disorders; Mental Disorder; Opioid
Keywords: Opiate treatment; Opioid treatment; Glucagon-Like Peptide-1 Agonist; Opioid use disorder; Semaglutide
MeSH Terms: conditions — Opioid-Related Disorders; Behavior, Addictive; Narcotic-Related Disorders; Substance-Related Disorders; Chemically-Induced Disorders; Mental Disorders | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Investigational group (Experimental): Participants randomized to semaglutide will be started at a low dose (0.25 mg once per week) which will be gradually increased weekly until 1.0 mg is reached at Week 4 of the intervention.
  Interventions: Drug: Semaglutide Pen Injector
- Control group (Placebo Comparator): Participants in the control group will have placebo administered once per week.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide Pen Injector — Semaglutide will be provided using an injection pen
  Other Names: Ozempic
  Arms: Investigational group
Drug: Placebo — Placebo will be a dry needle stick; no substances will be injected
  Other Names: Dry needle stick
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to learn if semaglutide can reduce illicit opioid use in adults in outpatient treatment for opioid use disorder, and who are receiving either buprenorphine or methadone maintenance treatment. The main question it aims to answer is:

• Does semaglutide increase the likelihood that participants will refrain from using illicit and nonprescribed opioids?

The investigators will compare semaglutide to a placebo (a needle prick that contains no drug) to see if semaglutide works to reduce use of illicit and nonprescribed opioids.

The participants will:

* Take semaglutide or a placebo every week for 12 weeks
* Visit the clinic every week for urine drug screening and pregnancy testing, vital signs, and to complete mental health and drug use questionnaires
* Complete smartphone surveys sent at set times during the study

DETAILED DESCRIPTION:
The purpose of this study is to determine whether 12 weeks of once-weekly treatment with the glucagon-like peptide-1 receptor (GLP-1R) agonist, semaglutide, will reduce illicit opioid use over a 19 week period (129-172 days) among individuals in outpatient treatment for opioid use disorder, and who are receiving either buprenorphine or methadone maintenance treatment (i.e., medication for opioid use disorder; MOUD). Following successful consent and initiation of screening, participants will complete a baseline evaluation and begin a baseline data collection period. If screened into the study, they will be randomly assigned to semaglutide or placebo control arms, in a 1:1 ratio using a permuted-block randomization algorithm stratified by site and MOUD, and begin a 1-week baseline period. Semaglutide (injector pen) or placebo will be administered as a subcutaneously (SC) once per week for 12 weeks, starting at a dose of 0.25 mg SC and advanced on a fixed-flexible dose schedule, based on tolerability, to a dose of 1.0 mg SC per week, or the maximum tolerated dose if less than 1.0 mg. Participants will receive study intervention in an outpatient setting for a total of 12 weeks. After the 12-week intervention, participants will discontinue semaglutide or placebo and be observed for an additional week (wash-out period). A final follow-up visit will then take place approximately 4 weeks after the washout visit (calculated as 18 weeks after Baseline/Treatment Visit 1).

During each study visit, participants will undergo urine drug screening and pregnancy testing, vital signs collection, and complete mental health and drug use questionnaires. Participants will also complete smartphone surveys sent at set times during the study. Blood samples will be collected at 2 of the visits (screening and the study week 14) and a physical examination and medical history collection will be done at the baseline visit.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years.
* Body mass index (BMI) > 18.
* Able and willing to provide informed consent prior to any study-related activities.
* Current diagnosis of Diagnostic and Statistical Manual Diploma in Social Medicine (DSM)-5 Opioid Use Disorder (OUD) as per the Mini International Neuropsychiatric Interview (MINI) or per the site clinic diagnosis. Patients are eligible if they have a MINI > 3 ("moderate" or "severe" in the "Specify If" box in the Substance Use Disorder (Non-Alcohol) module for the category of opiates).
* Currently receiving outpatient treatment for OUD and at least 2 weeks on buprenorphine (BUP) or 4 weeks on methadone at the study site and/or at an associated clinic at the time of enrollment.
* Have at least 1 urine test positive for opioids after 2 weeks on BUP or 4 weeks on methadone.
* Have positive self-reporting of opioid use after 2 weeks on BUP or 4 weeks on methadone.
* If anatomically capable of becoming pregnant and of childbearing age, is not pregnant (confirmed) or breastfeeding at the time of enrollment and agrees to use a medically accepted method of birth control or to abstain from sexual intercourse while in the study.
* Able to read and communicate in English to the level required to accept standard care and complete all study requirements.
* Able and willing to engage/adhere to the entirety of the study protocol (19 weeks).
* Not currently a prisoner.

Exclusion Criteria:

* Age < 18 or > 75 years.
* BMI <18.
* Individuals who are pregnant, planning pregnancy, breastfeeding, or unwilling to use adequate contraceptive measures.
* Current use of glucagon-like peptide 1 receptor (GLP-1R) agonist.
* History of angioedema, serious hypersensitivity reaction, or anaphylactic reaction to semaglutide or another GLP-1R agonist.
* Personal or family history of medullary thyroid carcinoma (MTC) or patients with multiple endocrine neoplasia syndrome Type 2 (MEN 2) or thyroid nodule.
* Type 1 diabetes or history of diabetic ketoacidosis.
* Type 2 diabetes mellitus or current use of a dipeptidyl peptidase-4 (DPP-4) inhibitor.
* Past 30-day use of Sincalide, Sulfonylureas, insulin and insulin products or other medications that may interact with semaglutide.
* Hypoglycemia on intake visit (blood glucose < 60 mg/dL).
* End-stage renal failure, on dialysis, or glomerular filtration rate (GFR) <30 mL/min per 1.73 square meters or previous renal transplant.
* End stage liver disease or previous liver transplant.
* Current or past diagnosis of pancreatitis, gastroparesis, or other severe gastrointestinal (GI) disease.
* Current or past diagnosis of gallbladder disease or gallstones.
* Serious cardiovascular disease within the past 6 months (e.g. uncontrolled hypertension, heart failure, significant cardiac arrhythmias, myocardial infarction, presence of angina pectoris, symptomatic coronary artery disease, deep vein thrombosis, pulmonary embolism, second- or third-degree heart block, mitral valve or aortic stenosis, hypertrophic cardiomyopathy, stroke).
* Severe co-occurring psychiatric disorder (e.g., bipolar disorder, psychotic disorder, schizophrenia), and/or history or evidence of organic brain disease or dementia that would compromise safety or compliance with the study protocol in the opinion of the site principal investigator (PI) and/or physician. As there is no specific scale that determines this, this will include the Site PI/physician determining if the potential participant shows consistency in decision making and if they are alert and oriented to time, date, day and location.
* Significant risk of suicide requiring a different/higher level of care, according to the clinical judgment of the study physician or site principal investigator, or history of suicide attempts within the past 1 year, unless participation is cleared by clinician assessment and/or judgment. A Columbia-Suicide Severity Rating Scale (C-SSRS) indicating a history of suicide attempts within the past year, or active suicidal ideation within the past 1 month, will qualify as significant risk of suicide.
* Treatment with any investigational drug in the one month preceding the study.
* Any contraindication to both methadone and BUP.
* Any contraindication to a GLP-1R agonist.
* Previous randomization for participation in this trial.
* Any other condition at screening that precludes safe participation in the trial in the judgment of the site PI or study physician.
* Plans for travel outside of the local area over the 19 weeks (1 week of baseline, 12 weeks of medication, 1 week wash-out, and follow-up after a further 28 days) that would interfere with visits during the study period or other logistic factors that would make it difficult to commit to the entire duration of study.
* Currently a prisoner.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants being abstinent from illicit and nonprescribed opioids. | Study week 2
  Each week in the 12 week trial period will be rated as abstinent if both urine test and participants' report by Timeline FollowBack (TLFB) questionnaire are negative for illicit/non-prescribed opioids, or urine is negative and TLFB missing, or TLFB negative and urine missing; and not abstinent otherwise (either urine positive, or TLFB positive, or both are missing). For certain opioids (e.g., fentanyl), declining rates in urine will be considered negative for usage.
Number of participants being abstinent from illicit and nonprescribed opioids. | Study week 3
  Each week in the 12 week trial period will be rated as abstinent if both urine test and participants' report by Timeline FollowBack (TLFB) questionnaire are negative for illicit/non-prescribed opioids, or urine is negative and TLFB missing, or TLFB negative and urine missing; and not abstinent otherwise (either urine positive, or TLFB positive, or both are missing). For certain opioids (e.g., fentanyl), declining rates in urine will be considered negative for usage.
Number of participants being abstinent from illicit and nonprescribed opioids. | Study week 4
  Each week in the 12 week trial period will be rated as abstinent if both urine test and participants' report by Timeline FollowBack (TLFB) questionnaire are negative for illicit/non-prescribed opioids, or urine is negative and TLFB missing, or TLFB negative and urine missing; and not abstinent otherwise (either urine positive, or TLFB positive, or both are missing). For certain opioids (e.g., fentanyl), declining rates in urine will be considered negative for usage.
Number of participants being abstinent from illicit and nonprescribed opioids. | Study week 5
  Each week in the 12 week trial period will be rated as abstinent if both urine test and participants' report by Timeline FollowBack (TLFB) questionnaire are negative for illicit/non-prescribed opioids, or urine is negative and TLFB missing, or TLFB negative and urine missing; and not abstinent otherwise (either urine positive, or TLFB positive, or both are missing). For certain opioids (e.g., fentanyl), declining rates in urine will be considered negative for usage.
Number of participants being abstinent from illicit and nonprescribed opioids. | Study week 6
  Each week in the 12 week trial period will be rated as abstinent if both urine test and participants' report by Timeline FollowBack (TLFB) questionnaire are negative for illicit/non-prescribed opioids, or urine is negative and TLFB missing, or TLFB negative and urine missing; and not abstinent otherwise (either urine positive, or TLFB positive, or both are missing). For certain opioids (e.g., fentanyl), declining rates in urine will be considered negative for usage.
Number of participants being abstinent from illicit and nonprescribed opioids. | Study week 7
  Each week in the 12 week trial period will be rated as abstinent if both urine test and participants' report by Timeline FollowBack (TLFB) questionnaire are negative for illicit/non-prescribed opioids, or urine is negative and TLFB missing, or TLFB negative and urine missing; and not abstinent otherwise (either urine positive, or TLFB positive, or both are missing). For certain opioids (e.g., fentanyl), declining rates in urine will be considered negative for usage.
Number of participants being abstinent from illicit and nonprescribed opioids. | Study week 8
  Each week in the 12 week trial period will be rated as abstinent if both urine test and participants' report by Timeline FollowBack (TLFB) questionnaire are negative for illicit/non-prescribed opioids, or urine is negative and TLFB missing, or TLFB negative and urine missing; and not abstinent otherwise (either urine positive, or TLFB positive, or both are missing). For certain opioids (e.g., fentanyl), declining rates in urine will be considered negative for usage.
Number of participants being abstinent from illicit and nonprescribed opioids. | Study week 9
  Each week in the 12 week trial period will be rated as abstinent if both urine test and participants' report by Timeline FollowBack (TLFB) questionnaire are negative for illicit/non-prescribed opioids, or urine is negative and TLFB missing, or TLFB negative and urine missing; and not abstinent otherwise (either urine positive, or TLFB positive, or both are missing). For certain opioids (e.g., fentanyl), declining rates in urine will be considered negative for usage.
Number of participants being abstinent from illicit and nonprescribed opioids. | Study week 10
  Each week in the 12 week trial period will be rated as abstinent if both urine test and participants' report by Timeline FollowBack (TLFB) questionnaire are negative for illicit/non-prescribed opioids, or urine is negative and TLFB missing, or TLFB negative and urine missing; and not abstinent otherwise (either urine positive, or TLFB positive, or both are missing). For certain opioids (e.g., fentanyl), declining rates in urine will be considered negative for usage.
Number of participants being abstinent from illicit and nonprescribed opioids. | Study week 11
  Each week in the 12 week trial period will be rated as abstinent if both urine test and participants' report by Timeline FollowBack (TLFB) questionnaire are negative for illicit/non-prescribed opioids, or urine is negative and TLFB missing, or TLFB negative and urine missing; and not abstinent otherwise (either urine positive, or TLFB positive, or both are missing). For certain opioids (e.g., fentanyl), declining rates in urine will be considered negative for usage.
Number of participants being abstinent from illicit and nonprescribed opioids. | Study week 12
  Each week in the 12 week trial period will be rated as abstinent if both urine test and participants' report by Timeline FollowBack (TLFB) questionnaire are negative for illicit/non-prescribed opioids, or urine is negative and TLFB missing, or TLFB negative and urine missing; and not abstinent otherwise (either urine positive, or TLFB positive, or both are missing). For certain opioids (e.g., fentanyl), declining rates in urine will be considered negative for usage.
Number of participants being abstinent from illicit and nonprescribed opioids. | Study week 13
  Each week in the 12 week trial period will be rated as abstinent if both urine test and participants' report by Timeline FollowBack (TLFB) questionnaire are negative for illicit/non-prescribed opioids, or urine is negative and TLFB missing, or TLFB negative and urine missing; and not abstinent otherwise (either urine positive, or TLFB positive, or both are missing). For certain opioids (e.g., fentanyl), declining rates in urine will be considered negative for usage.

SECONDARY OUTCOMES:
Self-reported opioid craving scores as assessed via smartphone surveys | Study week 1
  Validated 0-4 scale measuring desire/intention to use drug where 0 is no desire/intention and 4 is the highest desire/intention
Self-reported opioid craving scores as assessed via smartphone surveys | Study week 2
  Validated 0-4 scale measuring desire/intention to use drug where 0 is no desire/intention and 4 is the highest desire/intention
Self-reported opioid craving scores as assessed via smartphone surveys | Study week 5
  Validated 0-4 scale measuring desire/intention to use drug where 0 is no desire/intention and 4 is the highest desire/intention
Self-reported opioid craving scores as assessed via smartphone surveys | Study week 9
  Validated 0-4 scale measuring desire/intention to use drug where 0 is no desire/intention and 4 is the highest desire/intention
Self-reported opioid craving scores as assessed via smartphone surveys | Study week 13
  Validated 0-4 scale measuring desire/intention to use drug where 0 is no desire/intention and 4 is the highest desire/intention
Self-reported opioid craving scores as assessed via smartphone surveys | Study week 14
  Validated 0-4 scale measuring desire/intention to use drug where 0 is no desire/intention and 4 is the highest desire/intention
Self-reported opioid craving scores as assessed via smartphone surveys | Study week 18
  Validated 0-4 scale measuring desire/intention to use drug where 0 is no desire/intention and 4 is the highest desire/intention
Self-reported opioid craving as assessed via In-person Cravings Scales scores | Study week 2
  Validated 0-4 scale measuring desire/intention to use drug where 0 is no desire/intention and 4 is the highest desire/intention
Self-reported opioid craving as assessed via In-person Cravings Scales scores | Study week 3
  Validated 0-4 scale measuring desire/intention to use drug where 0 is no desire/intention and 4 is the highest desire/intention
Self-reported opioid craving as assessed via In-person Cravings Scales scores | Study week 4
  Validated 0-4 scale measuring desire/intention to use drug where 0 is no desire/intention and 4 is the highest desire/intention
Self-reported opioid craving as assessed via In-person Cravings Scales scores | Study week 5
  Validated 0-4 scale measuring desire/intention to use drug where 0 is no desire/intention and 4 is the highest desire/intention
Self-reported opioid craving as assessed via In-person Cravings Scales scores | Study week 6
  Validated 0-4 scale measuring desire/intention to use drug where 0 is no desire/intention and 4 is the highest desire/intention
Self-reported opioid craving as assessed via In-person Cravings Scales scores | Study week 7
  Validated 0-4 scale measuring desire/intention to use drug where 0 is no desire/intention and 4 is the highest desire/intention
Self-reported opioid craving as assessed via In-person Cravings Scales scores | Study week 8
  Validated 0-4 scale measuring desire/intention to use drug where 0 is no desire/intention and 4 is the highest desire/intention
Self-reported opioid craving as assessed via In-person Cravings Scales scores | Study week 9
  Validated 0-4 scale measuring desire/intention to use drug where 0 is no desire/intention and 4 is the highest desire/intention
Self-reported opioid craving as assessed via In-person Cravings Scales scores | Study week 10
  Validated 0-4 scale measuring desire/intention to use drug where 0 is no desire/intention and 4 is the highest desire/intention
Self-reported opioid craving as assessed via In-person Cravings Scales scores | Study week 11
  Validated 0-4 scale measuring desire/intention to use drug where 0 is no desire/intention and 4 is the highest desire/intention
Self-reported opioid craving as assessed via In-person Cravings Scales scores | Study week 12
  Validated 0-4 scale measuring desire/intention to use drug where 0 is no desire/intention and 4 is the highest desire/intention
Self-reported opioid craving as assessed via In-person Cravings Scales scores | Study week 13
  Validated 0-4 scale measuring desire/intention to use drug where 0 is no desire/intention and 4 is the highest desire/intention
Number of subjects who sustained abstinence from opioids (Binary indicator) | Study week 10
  Weekly abstinence rating (see primary outcome above) is rated as abstinent over the last 4 weeks for the treatment period.
Number of subjects who sustained abstinence from opioids (Binary indicator) | Study week 11
  Weekly abstinence rating (see primary outcome above) is rated as abstinent over the last 4 weeks for the treatment period.
Number of subjects who sustained abstinence from opioids (Binary indicator) | Study week 12
  Weekly abstinence rating (see primary outcome above) is rated as abstinent over the last 4 weeks for the treatment period.
Number of subjects who sustained abstinence from opioids (Binary indicator) | Study week 13
  Weekly abstinence rating (see primary outcome above) is rated as abstinent over the last 4 weeks for the treatment period.
Number of subjects abstinent from stimulants (i.e. cocaine or non-prescribed amphetamines) (Binary indicator) | Study week 10
  Weekly abstinence rating (see primary outcome above) is rated as abstinent over the last 4 weeks for the treatment period.
Number of subjects abstinent from stimulants (i.e. cocaine or non-prescribed amphetamines) (Binary indicator) | Study week 11
  Weekly abstinence rating (see primary outcome above) is rated as abstinent over the last 4 weeks for the treatment period.
Number of subjects abstinent from stimulants (i.e. cocaine or non-prescribed amphetamines) (Binary indicator) | Study week 12
  Weekly abstinence rating (see primary outcome above) is rated as abstinent over the last 4 weeks for the treatment period.
Number of subjects abstinent from stimulants (i.e. cocaine or non-prescribed amphetamines) (Binary indicator) | Study week 13
  Weekly abstinence rating (see primary outcome above) is rated as abstinent over the last 4 weeks for the treatment period.
Days using stimulants over the 12-week treatment period by Timeline Followback questionnaire | Study week 2
  Validated daily binary indicator for measuring use of stimulants
Days using stimulants over the 12-week treatment period by Timeline Followback questionnaire | Study week 3
  Validated daily binary indicator for measuring use of stimulants
Days using stimulants over the 12-week treatment period by Timeline Followback questionnaire | Study week 4
  Validated daily binary indicator for measuring use of stimulants
Days using stimulants over the 12-week treatment period by Timeline Followback questionnaire | Study week 5
  Validated daily binary indicator for measuring use of stimulants
Days using stimulants over the 12-week treatment period by Timeline Followback questionnaire | Study week 6
  Validated daily binary indicator for measuring use of stimulants
Days using stimulants over the 12-week treatment period by Timeline Followback questionnaire | Study week 7
  Validated daily binary indicator for measuring use of stimulants
Days using stimulants over the 12-week treatment period by Timeline Followback questionnaire | Study week 8
  Validated daily binary indicator for measuring use of stimulants
Days using stimulants over the 12-week treatment period by Timeline Followback questionnaire | Study week 9
  Validated daily binary indicator for measuring use of stimulants
Days using stimulants over the 12-week treatment period by Timeline Followback questionnaire | Study week 10
  Validated daily binary indicator for measuring use of stimulants
Days using stimulants over the 12-week treatment period by Timeline Followback questionnaire | Study week 11
  Validated daily binary indicator for measuring use of stimulants
Days using stimulants over the 12-week treatment period by Timeline Followback questionnaire | Study week 12
  Validated daily binary indicator for measuring use of stimulants
Days using stimulants over the 12-week treatment period by Timeline Followback questionnaire | Study week 13
  Validated daily binary indicator for measuring use of stimulants
Days using opioids over the 12-week treatment period by Timeline Followback questionnaire | Study week 2
  Validated daily binary indicator for measuring use of opioids
Days using opioids over the 12-week treatment period by Timeline Followback questionnaire | Study week 3
  Validated daily binary indicator for measuring use of opioids
Days using opioids over the 12-week treatment period by Timeline Followback questionnaire | Study week 4
  Validated daily binary indicator for measuring use of opioids
Days using opioids over the 12-week treatment period by Timeline Followback questionnaire | Study week 5
  Validated daily binary indicator for measuring use of opioids
Days using opioids over the 12-week treatment period by Timeline Followback questionnaire | Study week 6
  Validated daily binary indicator for measuring use of opioids
Days using opioids over the 12-week treatment period by Timeline Followback questionnaire | Study week 7
  Validated daily binary indicator for measuring use of opioids
Days using opioids over the 12-week treatment period by Timeline Followback questionnaire | Study week 8
  Validated daily binary indicator for measuring use of opioids
Days using opioids over the 12-week treatment period by Timeline Followback questionnaire | Study week 9
  Validated daily binary indicator for measuring use of opioids
Days using opioids over the 12-week treatment period by Timeline Followback questionnaire | Study week 10
  Validated daily binary indicator for measuring use of opioids
Days using opioids over the 12-week treatment period by Timeline Followback questionnaire | Study week 11
  Validated daily binary indicator for measuring use of opioids
Days using opioids over the 12-week treatment period by Timeline Followback questionnaire | Study week 12
  Validated daily binary indicator for measuring use of opioids
Days using opioids over the 12-week treatment period by Timeline Followback questionnaire | Study week 13
  Validated daily binary indicator for measuring use of opioids

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Nyland, PhD, Principal Investigator — Milton S. Hershey Medical Center
Locations (3):
- United States (3):
  - University of Maryland Baltimore, Baltimore, Maryland
  - NYU Langone Health, New York, New York
  - Pennsylvania Psychiatric Institute, Harrisburg, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Only summary data will be made available. No individual participant data (IPD) will be shared with other researchers.

REFERENCES:
- [Derived] Freet CS, Shuler K, Kawasaki S, Weintraub E, Greenblatt A, Kladney M, Nunes E, Foster KL, Kong L, Raja-Khan N, Cleveland HH, Grigson PS, Bunce SC, Brick TR, Nyland JE. Efficacy of the GLP-1 receptor agonist, semaglutide, in abstinence from illicit and nonprescribed opioids in an outpatient population with OUD: a randomized, double-blind, placebo-controlled clinical trial protocol. Addict Sci Clin Pract. 2025 Oct 30;20(1):89. doi: 10.1186/s13722-025-00618-2. PMID 41168808
- [Derived] Freet CS, Shuler K, Kawasaki S, Weintraub E, Greenblatt A, Kladney M, Nunes E, Foster KL, Kong L, Raja-Khan N, Cleveland HH, Grigson PS, Bunce SC, Brick TR, Nyland JE. Efficacy of the GLP-1 receptor agonist, semaglutide, in abstinence from illicit and nonprescribed opioids in an outpatient population with treatment-refractory OUD: A randomized, double-blind, placebo-controlled clinical trial protocol. Res Sq [Preprint]. 2025 May 26:rs.3.rs-6666196. doi: 10.21203/rs.3.rs-6666196/v1. PMID 40502777